CLINICAL TRIAL: NCT06943287
Title: A Remote Pharmacist Intervention to Improve Smoking Cessation
Brief Title: Pharmacist Intervention to Improve Smoking Cessation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Jacob E. Simmering, Assistant Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202411248
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist Intervention Group (Experimental)
  Interventions: Behavioral: Pharmacist Intervention
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Pharmacist Intervention — If the patient is randomized to the intervention group, they will complete a series of phone calls with the research pharmacist. These will occur at baseline (within 1 to 2 days of enrollment), 2-weeks, 4-weeks, 6-weeks, 8-weeks, 10-weeks, and 12-weeks. During these calls, the research pharmacist will ask the patient about any past quit attempts; when they had their last cigarette; if they have been prescribed any cessation medications; if they have picked up their medication; if they have started the medication; they will assess their stage of change for quitting; discuss pros, cons, and barriers of quitting; behavioral responses to triggers/urges; and make any necessary nicotine replacement therapy (NRT; i.e., nicotine patches, gums, lozenges, inhalers, and/or nasal sprays) changes. Each call is expected to take 20-30 minutes.
  Arms: Pharmacist Intervention Group

SUMMARY:
The goal of this study is to assess the effectiveness of a remote pharmacist intervention to help smokers quit.

The main questions it aims to answer are:

* Will smokers being screened for lung cancer with low-radiation-level chest computed tomography (CT) be willing to participate in this study and talk to the pharmacist about smoking cessation?
* Will those in the intervention group be more likely to report smoking cessation than those in the control group.

Participants in the intervention group will be asked to complete a baseline survey; speak with a pharmacist via phone call at baseline, 2 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, and 12 weeks; and complete an exit survey.

Participants in the control group will be asked to complete a baseline survey and an exit survey.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker
* Current patient in the Lung Cancer Screening Program

Exclusion Criteria:

* Unable to speak/read English
* Unable to provide their own written informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of Interactions with Pharmacist | 12 weeks
  The number of phone calls the intervention participants complete with the research pharmacist.

SECONDARY OUTCOMES:
Number of Nicotine Replacement Therapies Used to Quit Smoking | 12 weeks
  The number of participants who use nicotine replacement therapies during the study.
Number of Non-Medication Tool Used to Quit Smoking | 12 weeks
  The number of participants who use non-medication tools to quit smoking.
Number of Successful Quit Attempts | 12 weeks
  The number of participants who have successfully quit smoking at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob E Simmering, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Health Care, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No